CLINICAL TRIAL: NCT03832608
Title: Relationship Between the Sarcopenia Diagnostic Cut-points and Functionality in Older Adults
Brief Title: Sarcopenia Cut-points and Functionality in Older Adults
Acronym: SARCOFUNC
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Maria dels Angels Cebria i Iranzo, PT, PhD, Assistant professor, University of Valencia
Other Study IDs: H1542733812827; H1542733812827 (Other: University of Valencia Research Ethics Committee)
Record Dates: First submitted 2019-01-31; First posted 2019-02-06 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Sarcopenia; Diagnostic
Keywords: Older adult; Sarcopenia; Frailty; Functionality; Muscle strength; Muscle mass; Walk speed
MeSH Terms: conditions — Sarcopenia; Disease; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Older adults and Sarcopenia: Older adults with and without Sarcopenia living in Valencia Province.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is not intervention to be administered, only collection of data through various tests and questionnaires.

SUMMARY:
This is a cross-sectional study conducted in older adults living in Valencia Province in order to establish the cut-off points of the multicriteria diagnostic of sarcopenia through functionality and frailty variables.

DETAILED DESCRIPTION:
Sarcopenia is a geriatric syndrome that involves a gradual and generalized loss of the mass and strength of the skeletal muscles. Currently, there is an international debate about the criteria and reference values for the sarcopenia diagnosis, and the main scientific societies encourage improving research on this. The biggest problem lies in the assessment of the diagnostic criterion of muscle mass while the criterion of muscular strength seems safer and more robust. Experts point out the need to adjust the muscle mass indexes to the characteristics of the population studied, and the convenience of relating the three diagnostic criteria of sarcopenia (muscle mass and strength, and walking speed) with other variables that report about functionality and frailty in older adults.

The main objective is to establish different cut-off points for the diagnostic criteria of sarcopenia and relate them with other instruments for assessing functionality in older population of Valencia Province.

To this purpose, data will be collected through various tests and questionnaires about: clinical, demographic and anthropometric characteristics; muscle mass; muscle strength; walk speed; physical and cognitive function; nutritional status; self-perception of health; comorbidity and frailty. With this information it will be possible, as primary outcome, to determine a more sensitive, reliable and valid muscle mass index to predict sarcopenia, and, as a secondary outcome, to establish the relationship between the multicriteria diagnostic of sarcopenia with the functional and frailty variables.

ELIGIBILITY:
Inclusion Criteria:

* People aged > 65 years
* Residents in Valencia Province (Living-Community, Day-Centers and institutionalized)

Exclusion Criteria:

* Lobo Mini-exam cognoscitive < 18 score
* Any disorder that prevents from performing the assessment tests.
* Recent hospitalization or who are in a acute process of any illness (less one month).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults (+65 years) living in Valence Province.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
First criteria of sarcopenia diagnostic: hand grip strength | The cohort group will be assessed in one day visit.
  Muscle strength measured by the isometric hand grip strength (reference: Age and Aging. 2010;39:412-23).
First criteria of sarcopenia diagnostic: knew extension strength | The cohort group will be assessed in one day visit.
  Muscle strength measured by the isometric knew extension (reference: Phys Ther. 1996;76(3):248-59).
First criteria of sarcopenia diagnostic: elbow flexion strength | The cohort group will be assessed in one day visit.
  Muscle strength measured by the isometric elbow flexion (reference: Phys Ther. 1996;76(3):248-59).
Second criteria of sarcopenia diagnostic: muscle mass | The cohort group will be assessed in one day visit.
  Muscle mass estimated by Bioimpedance analysis (BIA) (reference: J Aging Phys Act. 2015;23(4):597-606).
Third criteria of sarcopenia diagnostic: walk speed | The cohort group will be assessed in one day visit.
  Walk speed measured by the Short Physical Performance Balance test (SPPB) (reference: J Gerontol A Biol Sci Med Sc 2000; 55(4):M221-31.

SECONDARY OUTCOMES:
Functionality: Modified Baecke Questionnaire | The cohort group will be assessed in one day visit.
  Functionality measured by the Modified Baecke Questionnaire (reference: Med Clin.2007;129:326-32). The Modified Baecke Questionnaire results in a score to classify people as high, moderate, or low in daily physical activity, based on tertiles.
  Work Index = 0 1 +12 + 13 + 14 + 15 + 16 + 17 + I8)/8 Sport Index = 0 9 + 110 + II1 + I12)/4 Leisure Time Index = 0 ' 3 + 114 + 115 + 116 + 117 + 118 + I19V7 Total Index = work index + sports index + leisure time index.
Functionality: Barthel Index | The cohort group will be assessed in one day visit.
  Functionality measured by the Barthel Index (reference: Rev Esp Geriatr Gerontol.1993;28:32-40). Range from 0 to 100 score. High score of 100 means total independent.
Functionality: Lawton and Brody Questionnaire | The cohort group will be assessed in one day visit.
  Functionality measured by the Lawton and Brody Questionnaire (reference: Gerontologist.1969;9:179-86).Range from 0 to 8 score. High score of 8 means total independent to perform daily activities.
Frailty: Fried Scale | The cohort group will be assessed in one day visit.
  Frailty measured by the Fried Scale (reference: J Gerontol A Biol Sci Med Sc. 2001;56(3):M146-56). It is a scale with 5 domains: weight loss, self-reported exhaustion, physical activity, walking speed, and weakness. It has a total score ≥ 5 points. A frail person is who scores 3 to 5; is prefrail when scores is 1 to 2, and robust if scores is 0.
Frailty:Frail Scale | The cohort group will be assessed in one day visit.
  Frailty measured by the Frail Scale (reference: J Nutr Health Aging. 2012;16(7):601-8). It has a total score of 5 points. The more score the more frailty. As in Fried scale, participants with scores 3 to 5 is frail person; with scores 1 to 2 is prefrail, and robust if scores is 0.
Frailty: Kihon Check List (KCL) | The cohort group will be assessed in one day visit.
  Frailty measured by the Kihon Check List (reference: Geriatr Gerontol Int. 2016;16(6):709-15). The KCL is a simple self-reporting yes/no survey consisting of 25 questions structured into seven domains /dimensions. A total score ≥ 10 points allow to identify a frail person and each domain can identify the specific need.
Comorbidity | The cohort group will be assessed in one day visit.
  Comorbidity measured by Abbreviated Charslon Index (reference: J Chron Dis.1987;40:373-83). Range from 0 to 10 score. High score of 10 means high comorbidity; 0 means absence of comorbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Cebrià i Iranzo, PT, PhD, Principal Investigator — University of Valencia; Mercè Balasch i Bernat, PT, PhD, Study Chair — University of Valencia; Anna Arnal Gómez, PT, PhD, Study Chair — University of Valencia; Trinidad Sentandreu Mañó, PT, PhD, Study Chair — University of Valencia; Maria A Tortosa Chuliá, PhD, Study Chair — University of Valencia; Natalia Cezón Serrano, PT, Study Chair — University of Valencia; Jose M Tomás, PhD, Study Chair — University of Valencia; Silvia Forcano Sanjuán, MD, Study Chair — Hospital Universitari i Politècnic La Fe (Valencia)
Locations (1):
- Armonea Group, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Masanes F, Culla A, Navarro-Gonzalez M, Navarro-Lopez M, Sacanella E, Torres B, Lopez-Soto A. Prevalence of sarcopenia in healthy community-dwelling elderly in an urban area of Barcelona (Spain). J Nutr Health Aging. 2012 Feb;16(2):184-7. doi: 10.1007/s12603-011-0108-3. PMID 22323356
- [Background] Salva A, Serra-Rexach JA, Artaza I, Formiga F, Rojano I Luque X, Cuesta F, Lopez-Soto A, Masanes F, Ruiz D, Cruz-Jentoft AJ. [Prevalence of sarcopenia in Spanish nursing homes: Comparison of the results of the ELLI study with other populations]. Rev Esp Geriatr Gerontol. 2016 Sep-Oct;51(5):260-4. doi: 10.1016/j.regg.2016.02.004. Epub 2016 Apr 9. Spanish. PMID 27068239
- [Background] Chen LK, Liu LK, Woo J, Assantachai P, Auyeung TW, Bahyah KS, Chou MY, Chen LY, Hsu PS, Krairit O, Lee JS, Lee WJ, Lee Y, Liang CK, Limpawattana P, Lin CS, Peng LN, Satake S, Suzuki T, Won CW, Wu CH, Wu SN, Zhang T, Zeng P, Akishita M, Arai H. Sarcopenia in Asia: consensus report of the Asian Working Group for Sarcopenia. J Am Med Dir Assoc. 2014 Feb;15(2):95-101. doi: 10.1016/j.jamda.2013.11.025. PMID 24461239
- [Background] Lee WJ, Liu LK, Peng LN, Lin MH, Chen LK; ILAS Research Group. Comparisons of sarcopenia defined by IWGS and EWGSOP criteria among older people: results from the I-Lan longitudinal aging study. J Am Med Dir Assoc. 2013 Jul;14(7):528.e1-7. doi: 10.1016/j.jamda.2013.03.019. Epub 2013 May 10. PMID 23664768
- [Background] Ethgen O, Beaudart C, Buckinx F, Bruyere O, Reginster JY. The Future Prevalence of Sarcopenia in Europe: A Claim for Public Health Action. Calcif Tissue Int. 2017 Mar;100(3):229-234. doi: 10.1007/s00223-016-0220-9. Epub 2016 Dec 24. PMID 28012107
- [Result] Cebria I Iranzo MA, Arnal-Gomez A, Tortosa-Chulia MA, Balasch-Bernat M, Forcano S, Sentandreu-Mano T, Tomas JM, Cezon-Serrano N. Functional and Clinical Characteristics for Predicting Sarcopenia in Institutionalised Older Adults: Identifying Tools for Clinical Screening. Int J Environ Res Public Health. 2020 Jun 22;17(12):4483. doi: 10.3390/ijerph17124483. PMID 32580427
- [Result] Arnal-Gomez A, Cebria I Iranzo MA, Tomas JM, Tortosa-Chulia MA, Balasch-Bernat M, Sentandreu-Mano T, Forcano S, Cezon-Serrano N. Using the Updated EWGSOP2 Definition in Diagnosing Sarcopenia in Spanish Older Adults: Clinical Approach. J Clin Med. 2021 Mar 2;10(5):1018. doi: 10.3390/jcm10051018. PMID 33801427
- [Derived] Balasch-Bernat M, Sentandreu-Mano T, Tomas JM, Cebria I Iranzo MA, Tortosa-Chulia MA, Arnal-Gomez A, Cezon-Serrano N. Deepening the understanding of the structural validity of the Tilburg Frailty Indicator. Aging Clin Exp Res. 2023 Jun;35(6):1263-1271. doi: 10.1007/s40520-023-02407-w. Epub 2023 Apr 21. PMID 37085651